CLINICAL TRIAL: NCT05900115
Title: The Middle Years Study: A Feasibility Study of a Self-paced Program Designed to Provide Parents of Middle School-aged Students With Knowledge About Teen Substance Use and Practice in High Quality Parent-adolescent Communication Methods Delivered Through a Highly Interactive Web-based Software Application
Brief Title: Feasibility Study of a Web-based Program to Help Parents of Middle School Students Effectively Communicate With Their Children About Substance Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MiddleYearsStudyR21-23-003-001; 5R21DA052737-02 (NIH)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Substance Use; Parenting; Communication
MeSH Terms: conditions — Substance-Related Disorders; Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be informed which condition they are assigned (intervention or active control). All measures are assessed using a web-based data collection system rather than a human outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based intervention (Experimental): The intervention is a web-based resource that provides parents with media literacy and media mediation skills, knowledge about adolescent development and substance use, and practice in high quality parent-child communication.
  Interventions: Behavioral: Media Ready Parent
- Active Control Program (Active Comparator): The active control is a web-based resource that contains PDFs of medically accurate information about adolescent substance use.
  Interventions: Behavioral: Active Control Program

INTERVENTIONS:
Behavioral: Media Ready Parent — The intervention is a web-based resource that provides parents with media literacy and media mediation skills, knowledge about adolescent development and substance use, and practice in high quality parent-child communication.
  Arms: Web-based intervention
Behavioral: Active Control Program — The active control is a web-based resource that contains PDFs of medically accurate information about adolescent substance use.
  Arms: Active Control Program

SUMMARY:
The goal of this study is to test the feasibility of a web-based program for parents of middle school aged students. 286 parents and their child in 6th, 7th, or 8th grade will be asked to each complete two online questionnaires over the course of about a month, parents will also complete a web-based program between questionnaires. Researchers will compare the intervention and an active control to test the intervention program efficacy for improving outcomes related to parent-child communication, media message processing, and adolescent health.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and assess a self-administered, web-based program designed to increase parent knowledge about adolescent substance use, active media mediation skills, and practice high-quality parent-adolescent communication methods. The program will help parents of middle-school aged students, 6th-8th graders, communicate effectively about substance use and enhance media literacy skills to counter unhealthy media messages. Prevention efforts are most impacting for adolescents in middle school years as this is the time frame for growing independence, desire to fit-in and an increase risk for their own experimentation with substances.

ELIGIBILITY:
Inclusion Criteria:

* The adult must be the legal guardian of a child in 6th, 7th or 8th grade (known hereafter as "parent").
* The parent must be able and willing to receive email and text communication as part of the study.
* The parent-child pair must have access to a smartphone with internet connection as the resource review will be completed online in a format that is best viewed on a smartphone.
* The parent-child pair must be fluent in English as the study materials are conducted in English.
* The parent must indicate that they will give the child participant privacy to complete the questionnaires
* Both the adult and child must agree to participate.

Exclusion Criteria:

* In an effort to ensure diversity in parent gender and race/ethnicity, not all eligible pairs who are interested in participating will be enrolled in the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- innovation Research and Training, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants in the Participant Flow data table represent the number of individual participants.
Period: Overall Study
Arm/Group | Web-based Intervention | Active Control Program
Started | 304 | 272
Completed Pretest | 206 | 188
Completed | 175 | 174
Not Completed | 129 | 98
Not completed — Lost to Follow-up | 129 | 98

BASELINE CHARACTERISTICS:
Population: Intervention group included 206 participants (103 parents and 103 children). The control group included 188 participants (94 parents and 94 children).
Groups:
- Total: Total of all reporting groups
Arm/Group | Web-based Intervention | Active Control Program | Total
Number analyzed (Participants) | 206 | 188 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Intervention group included 206 participants (103 parents and 103 children). The control group included 188 participants (94 parents and 94 children).
  years
    Parent: number analyzed (Participants) | 103 | 94 | 197
    Parent | 43.19 (7.26) | 40.85 (6.76) | 42.08 (7.11)
    Child: number analyzed (Participants) | 103 | 94 | 197
    Child | 12.64 (1.14) | 12.66 (1.36) | 12.65 (1.24)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Intervention group included 206 participants (103 parents and 103 children). The control group included 188 participants (94 parents and 94 children).
  Participants
    Parent: number analyzed (Participants) | 103 | 94 | 197
    Parent: Woman/Girl | 52 | 52 | 104
    Parent: Man/Boy | 50 | 41 | 91
    Parent: Nonbinary | 1 | 1 | 2
    Parent: Missing | 0 | 0 | 0
    Child: number analyzed (Participants) | 103 | 94 | 197
    Child: Woman/Girl | 46 | 43 | 89
    Child: Man/Boy | 56 | 48 | 104
    Child: Nonbinary | 0 | 2 | 2
    Child: Missing | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intervention group included 206 participants (103 parents and 103 children). The control group included 188 participants (94 parents and 94 children).
  Participants
    Parent: number analyzed (Participants) | 103 | 94 | 197
    Parent: Hispanic or Latino | 13 | 10 | 23
    Parent: Not Hispanic or Latino | 82 | 78 | 160
    Parent: Unknown or Not Reported | 8 | 6 | 14
    Child: number analyzed (Participants) | 103 | 94 | 197
    Child: Hispanic or Latino | 25 | 19 | 44
    Child: Not Hispanic or Latino | 78 | 74 | 152
    Child: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intervention group included 206 participants (103 parents and 103 children). The control group included 188 participants (94 parents and 94 children).
  Participants
    Parent: number analyzed (Participants) | 103 | 94 | 197
    Parent: American Indian or Alaska Native | 0 | 0 | 0
    Parent: Asian | 2 | 2 | 4
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 20 | 14 | 34
    Parent: White | 69 | 65 | 134
    Parent: More than one race | 3 | 5 | 8
    Parent: Unknown or Not Reported | 9 | 8 | 17
    Child: number analyzed (Participants) | 103 | 94 | 197
    Child: American Indian or Alaska Native | 1 | 0 | 1
    Child: Asian | 3 | 2 | 5
    Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child: Black or African American | 15 | 14 | 29
    Child: White | 70 | 62 | 132
    Child: More than one race | 11 | 14 | 25
    Child: Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 206 | 188 | 394

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parent Report of Parent-child Communication Quality at Week 4
Description: Parent-child communication quality will be adapted from the 16-item Parent-Adolescent Communication Scale (PACS; Barnes & Olson, 1985; Prado et al., 2007; α = .85). Participants are asked to indicate on a 4-point scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) the extent to which they agree with a series of 16 statements (e.g., I can discuss my beliefs with my child without feeling embarrassed). Higher scores indicate a better outcome. Responses on the items were averaged together.
Time Frame: Baseline and Week 4
Population: If a participant was missing data for any independent or dependent variables, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 74 | 78
score on a scale | 3.12 (0.03) | 3.11 (0.03)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — To examine intervention effects on primary outcomes at posttest, we used linear regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect; p = 0.77, Regression, Linear; Slope = 0.01, Standard Error of Mean .04

2. Primary Outcome: Change From Baseline in Child Report of Parent-child Communication Quality at Week 4
Description: Parent-child communication quality will be adapted from the 16-item Parent-Adolescent Communication Scale (PACS; Barnes & Olson, 1985; Prado et al., 2007; α = .85). Participants are asked to indicate on a 4-point scale (1=strongly disagree; 2=disagree; 3=agree; 4=strongly agree) the extent to which they agree with a series of 16 statements (e.g., I can discuss my beliefs with my parent without feeling embarrassed). Higher scores indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 70 | 78
score on a scale | 2.97 (0.04) | 2.95 (0.04)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.78, Regression, Linear; Slope = 0.02, Standard Error of Mean 0.06

3. Primary Outcome: Change From Baseline in Parent Report of Parent-child Substance Use Communication Frequency at Week 4
Description: Parent-child communication behaviors about substance use will be assessed by asking a series of 5 questions to assess the frequency of parent-child communication about alcohol, tobacco, vaping, marijuana, and prescription drugs (e.g., How much have you talked with your child about alcohol use?; 5-point Likert-type scale ranging from 1=Never to 5=Extremely Much). Adapted from adapted from Miller-Day & Kam (2010). Higher values indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: If a participant was missing any data on any covariates, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 102 | 93
score on a scale | 4.00 (0.08) | 3.87 (0.09)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.28, Regression, Linear; Slope = 0.13, Standard Error of Mean 0.12

4. Primary Outcome: Change From Baseline in Child Report of Parent-child Substance Use Communication Frequency at Week 4
Description: Parent-child communication behaviors about substance use will be assessed by asking a series of 5 questions to assess the frequency of parent-child communication about alcohol, tobacco, vaping, marijuana, and prescription drugs (e.g., How much has your parent talked with you about alcohol use?; 5-point Likert-type scale ranging from 1=Never to 5=Extremely Much). Adapted from adapted from Miller-Day & Kam (2010). Higher values indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 70 | 78
score on a scale | 3.66 (0.09) | 3.60 (0.09)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.68, Regression, Linear; Slope = 0.05, Standard Error of Mean 0.13

5. Primary Outcome: Change From Baseline in Parent Report of Parental Active Media Mediation at Week 4
Description: Parents' use of active media mediation strategies will be assessed using an adapted version of the Perceived Parental Media Mediation Scale (Valkenberg et al., 2013). The scale consists of four items (e.g., How often do you tell your child that what they see in media (like movies/TV, commercials, social media, and online content like YouTube) is different than real life?) measured on a 5-point Likert-type scale (1=Never; 2=almost never; 3=sometimes; 4=often; 5=very often). Higher scores indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: If a participant was missing any data on any covariates, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 102 | 93
score on a scale | 3.74 (0.09) | 3.42 (0.09)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.01, Regression, Linear; Slope = 0.32, Standard Error of Mean 0.13

6. Primary Outcome: Change From Baseline in Child Report of Parental Active Media Mediation at Week 4
Description: Child report of parent's use of active media mediation strategies will be assessed using an adapted version of the Perceived Parental Media Mediation Scale (Valkenberg et al., 2013). Child report of parent use of active media mediation strategies will be assessed using an adapted version of the Perceived Parental Media Mediation Scale (Valkenberg et al., 2013). The scale consists of four items (e.g., How often do your parents tell you that what they see in media (like movies/TV, commercials, social media, and online content like YouTube) is different than real life?) measured on a 5-point Likert-type scale (1=Never; 2=almost never; 3=sometimes; 4=often; 5=very often). Higher scores indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: If a participant was missing any data on any covariates, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 102 | 93
score on a scale | 3.27 (0.10) | 3.46 (0.10)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.18, Regression, Linear; Slope = -0.19, Standard Error of Mean 0.14

7. Primary Outcome: Change From Baseline in Parent Report of Parental Restrictive Media Mediation at Week 4
Description: Parents' use of restrictive media mediation strategies will be assessed using an adapted version of the Perceived Parental Media Mediation Scale (Valkenberg et al., 2013).The scale consists of four items (e.g., How often do you limit the amount of your child's screen time (watching shows, going online, playing video games, or using social media?) measured on a 5-point Likert-type scale (1=never; 2=almost never; 3=sometimes; 4=often; 5=very often). Higher scores indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: If a participant was missing any data on any covariates, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 102 | 93
score on a scale | 3.38 (0.08) | 3.36 (0.08)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.83, Regression, Linear; Slope = 0.03, Standard Error of Mean 0.12

8. Primary Outcome: Change From Baseline in Child Report of Parental Restrictive Media Mediation at Week 4
Description: Child report of parent's use of restrictive media mediation strategies will be assessed using an adapted version of the Perceived Parental Media Mediation Scale (Valkenberg et al., 2013). The scale consists of four items (e.g., How often do your parents tell you that you are not allowed to watch certain TV shows or movies because they are meant for adults?) measured on a 5-point Likert-type scale (1=never; 2=almost never; 3=sometimes; 4=often; 5=very often). Higher scores indicate a better outcome. Responses were averaged together.
Time Frame: Baseline and Week 4
Population: If a participant was missing any data on any covariates, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 102 | 93
score on a scale | 3.15 (0.09) | 3.23 (0.09)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.56, Regression, Linear; Slope = -.08, Standard Error of Mean 0.13

9. Primary Outcome: Change From Baseline in Child Substance Use Intentions at Week 4
Description: Substance use intentions will be assessed by asking "During the next year, do you think you will drink alcohol" (4-point scale; 1=I definitely will not; 2=I probably will not; 3=I probably will; 4=I definitely will; higher scores indicate a worse outcome). Questions will also be asked for use of tobacco, vape, marijuana, and prescription drugs without a prescription, for a total of 5 questions. Responses were averaged together and then dichotomized. Any participant with a mean of one ("I definitely will not") was rescored as "0" (no intentions) and any participant with a mean greater than one was rescored as "1" (any intentions). A rescored value of "1" indicated a worse outcome. Outcome measure type ("number") indicates the percentage of people who had a rescored value of "1" ("any intentions").
Time Frame: Baseline and Week 4
Population: Analyses were conducted using observed data instead of imputed.
Measure: Number; unit: percentage of participants with "1"
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 71 | 78
percentage of participants with "1" | 22.54 | 29.49
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — To examine intervention effects on primary dichotomous outcomes at posttest, we used logistic regression in intent-to-treat analyses. Posttest scores were regressed onto pretest scores, covariates, and the treatment effect; p = 0.85, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [.38 to 3.20], Standard Error of Mean .54

10. Primary Outcome: Change From Baseline in Child Willingness to Use Substances at Week 4
Description: Willingness to use substances will be assessed by asking "Suppose you were with a group of kids and they were drinking alcohol. How willing would you be to have a drink?" (4-point scale; 1=very unwilling; 2=unwilling; 3=willing; 4=very willing). Questions will also be asked for smoking, vaping, marijuana, and taking prescription drugs without a prescription. A total of 5 question will be asked, one for each substance type. Higher scores indicate a worse outcome. Responses were averaged.
Time Frame: Baseline and Week 4
Population: If a participant was missing any data on any covariates, they were not included in the outcome analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Web-based Intervention | Active Control Program
Number analyzed (Participants) | 102 | 93
score on a scale | 1.26 (.04) | 1.26 (.04)
Statistical Analysis 1: Comparison: Web-based Intervention vs Active Control Program; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 1.00, Regression, Linear; Slope = 0.00, Standard Error of Mean 0.05

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from pretest to posttest completion: approximately 4 weeks.
Arm/Group | Web-based Intervention | Active Control Program
All-Cause Mortality (participants affected / at risk) | 0/304 | 0/272
Serious Adverse Events (participants affected / at risk) | 0/304 | 0/272
Other Adverse Events (participants affected / at risk) | 0/304 | 0/272

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT05900115/Prot_SAP_000.pdf